CLINICAL TRIAL: NCT00685295
Title: Fentanyl Administered Intraorally for Rapid Treatment of Orthopedic Pain in the ED
Brief Title: Fentanyl Administered Intraorally for Rapid Treatment of Orthopedic Pain
Acronym: FAIRTOP
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Stephen H. Thomas, MD MPH, Attending Physician, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FAIRTOP
Record Dates: First submitted 2008-05-23; First posted 2008-05-28 (Estimated); Results first posted 2017-02-09 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2016-12

CONDITIONS: Pain, Fracture, Sprain
Keywords: Emergency Department; acute
MeSH Terms: conditions — Pain; Fractures, Bone; Sprains and Strains; Emergencies | interventions — Fentanyl; Lansoprazole; Oxycodone; oxycodone-acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 / Fentora (Experimental): Intervention Group:
  Subject receives:
  1. placebo oral/swallowed pill
  2. Fentanyl (Fentora) 100mcg rapidly dissolving transbuccal tablet
  Interventions: Drug: Fentanyl
- Arm 2 / Percocet/Prevacid (Active Comparator): Active Comparator Group:
  Subject receives:
  1. Oxycodone/APAP (Percocet) 5/325 mg oral/swallowed pill
  2. Lansoprazole 15 mg (Prevacid) comparator rapidly dissolving transbuccal tablet
  Interventions: Drug: Lansoprazole; Drug: Oxycodone

INTERVENTIONS:
Drug: Fentanyl — Fentanyl rapid dissolving tablet 100mcg
  Other Names: Fentora
  Arms: Arm 1 / Fentora
Drug: Lansoprazole — lansoprazole 15mg rapidly dissolving tablet
  Other Names: Prevacid SoluTab
  Arms: Arm 2 / Percocet/Prevacid
Drug: Oxycodone — Oxycodone 5/325 mg tablet
  Other Names: Percocet
  Arms: Arm 2 / Percocet/Prevacid

SUMMARY:
Assess whether transbuccal fentanyl provides more rapid relief of orthopedic pain, than does the comparator Percocet

DETAILED DESCRIPTION:
Patients will be initially deemed eligible for study consideration if, after MGH ED nursing triage, an X-ray is ordered for suspected isolated extremity injury and the triage acuity level is "Minor". Study staff (physicians) will monitor the ED registration and triage areas to assess whether triaged patients are potentially eligible.

For ED patients with minor isolated injuries, X-rays are often ordered from triage, where there is a supervising physician (or nurse practitioner) available to examine patients and direct care. Either at triage (for patients undergoing care at that location) or when patients are moved to the ED's Minor Surgery area, the supervising healthcare provider will be approached immediately after that individual's evaluation of the patient, and before any pain medication is administered, to begin the process of eligibility ascertainment.

If the provider agrees that the patient may be a candidate for the study, the next step will be for the provider to ask the patient if study staff may approach to discuss the trial.

If the patient agrees to have study staff approach to discuss the trial, study personnel (all EM resident or Attending-level physicians) will be introduced by healthcare providers to potential subjects. Study staff will then converse with the patients about the study's aims, methodology, and risks, confirming eligibility and determining if patients will consent to participate.

Patients who are approached, but who are determined to be ineligible, will have no data recorded, other than their age and race/ethnicity and the reason they were ineligible.

If eligible patients provide written consent in the manner and form dictated by Partners guidelines, the study procedures will commence.

For eligible patients who do not give consent, study physicians will emphasize that patient care will be unaffected by their decision. No further contact will occur between study staff and those patients. No identifying information about such patients will be recorded, but their age and race/ethnicity will be recorded. (Recording this information will allow for subsequent assessment for selection bias, and will also help search for patterns in patient types refusing analgesia trial participation.)

The actual medication administration will involve the following steps:

1. Patients participating in the study will be identified and placed in a "room" (stretcher or actual ED room) in the MGH ED's Minor Multipurpose (MIMP) area;
2. RNs will obtain the study medication pairs (buccal tablet + oral tablet) from the computerized medication storage area - RNs will take the next-numbered medication pair from the MGH Research Pharmacy-prepared drug packaging;
3. Actual medications will be administered by a licensed physician (a study co-investigator, EM resident or Attending physician at MGH), who is not the co-investigator monitoring the patient for endpoint assessment - the physician administering the medication/placebo will inform neither the patient nor the clinical or study staff, the identity of the medication/placebo pair given.

Patients will be monitored by a study physician co-investigator physically present with the patient, for a total of 120 minutes after administration of medication. They will be asked q-5-minutes, through 60 minutes, to rate their pain and degree of nausea, as well as to describe any adverse reactions to the medication. Both pain and nausea levels will be recorded using 10-point scales. Use of such scales is common in the pain literature, and is an emerging tool for evaluation of nausea.1,2 Data collection for analgesia efficacy will cease after 60 minutes, but patients will be monitored for at least another 60 minutes to maximize safety; patients will be assessed for discharge suitability by treating clinicians/nurses in the same fashion as other ED patients who receive opioids.

Vital signs (respiratory rate, blood pressure, heart rate, pulse oximetry) will be monitored for the two hours of the study. Continuous pulse oximetry will be used during the first study hour, and q5-minute spot-check pulse oximetry will be used during the second study hour; pulse oximetry monitoring will be changed to continuous mode during the second study hour if any spot-check reading falls below 98%. Other (non-pulse oximetry) vital signs will be monitored q5-minutes during the first study hour, and q15-minutes during the second study hour. These vital signs monitoring parameters represent the minimum for study subjects; treating clinicians or study staff physicians can increase the frequency of vital signs monitoring at their discretion. Any study subject not admitted to the hospital, will be discharged under the care of a responsible adult.

At the conclusion of the data collection period, patients will be asked if they would want to receive the same medication in the future. Other than a 24-hour telephone call (made only if patients agree), intended to assess for delayed problems such as nausea/vomiting, there will be no other study procedures or interventions.

ELIGIBILITY:
INCLUSION:

* 18-60 years of age
* Present to ED with a chief complaint of extremity injury
* Negative pregnancy test (urine or blood)
* Clinician judges subject to need extremity radiography to rule out a fracture
* Subjects must indicate that their pain is of sufficient severity to warrant treatment with a pain medication stronger than acetaminophen or aspirin.
* Subject's treating ED provider is aware of, and approves, participation (i.e. participation cannot be allowed to impair provision of standard patient care).

EXCLUSION:

* Treating provider judges that IV analgesia is required
* Allergy to acetaminophen or to any opiate/opioid
* Currently taking phenothiazines or CNS depressants (including alcohol), or if subject has taken MAO inhibitors or SSRIs within the past two weeks
* Already taken or been administered opioid analgesia for their current injury
* Chronic opioid therapy or if the subject (or their medical records) indicate a history of opioid abuse
* Breastfeeding mothers
* If subject is planning to drive home after their ED visit, or if they are judged for any other reason to be non-candidates for opioid therapy.
* hypersensitivity to lansoprazole
* phenylketonuria

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2008-08; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen H Thomas, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers.

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1 / Fentora: Subject receives placebo swallowed pill, and Fentora 100mcg rapidly dissolving transbuccal tablet
- Arm 2 / Percocet/Prevacid: Subject receives Percocet swallowed pill, and Prevacid comparator rapidly dissolving transbuccal tablet
Period: Overall Study
Arm/Group | Arm 1 / Fentora | Arm 2 / Percocet/Prevacid
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 / Fentora | Arm 2 / Percocet/Prevacid | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 30 | 60
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 29 (8) | 30 (12) | 30 (10)
Gender [Count of Participants; unit: Participants]
  Female | 10 | 12 | 22
  Male | 20 | 18 | 38
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 60.0

OUTCOME MEASURES:

1. Primary Outcome: Time to Analgesia
Description: Time it took for subjects to achieve a pain score reduction of 2 units (on a 0 to 10 scale)
Time Frame: 60 minutes
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Arm 1 / Fentora | Arm 2 / Percocet/Prevacid
Number analyzed (Participants) | 30 | 30
minutes | 10 [5 to 15] | 35 [20 to 40]

2. Primary Outcome: Pain Reduction
Description: Number of subjects who reached pain reduction. A subject was deemed to have reached pain reduction if there was a two-point drop in pain scale (0-10).
Time Frame: 60 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 / Fentora | Arm 2 / Percocet/Prevacid
Number analyzed (Participants) | 30 | 30
Participants | 30 | 24

3. Secondary Outcome: Occurrence of Untoward Opioid Side Effects
Description: Subjects were monitored for any signs of untoward opioid side effects.
Time Frame: 120 minutes
Measure: Count of Participants; unit: Participants
Groups:
- Arm 1 / Fentora: Intervention Group:
  Subject receives:
  1. placebo oral/swallowed pill
  2. Fentanyl (Fentora) 100mcg rapidly dissolving transbuccal tablet
  Fentanyl: Fentanyl rapid dissolving tablet 100mcg
- Arm 2 / Percocet/Prevacid: Active Comparator Group:
  Subject receives:
  1. Oxycodone/APAP (Percocet) 5/325 mg oral/swallowed pill
  2. Lansoprazole 15 mg (Prevacid) comparator rapidly dissolving transbuccal tablet
  Lansoprazole: lansoprazole 15mg rapidly dissolving tablet
  Oxycodone: Oxycodone 5/325 mg tablet
Arm/Group | Arm 1 / Fentora | Arm 2 / Percocet/Prevacid
Number analyzed (Participants) | 30 | 30
Participants | 0 | 1

ADVERSE EVENTS:
Time Frame: 1 day after enrollment, subjects were contacted
Arm/Group | Arm 1 / Fentora | Arm 2 / Percocet/Prevacid
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes